CLINICAL TRIAL: NCT04840875
Title: Phase I Clinical Trial of Autologous CD7-CAR T Cells in the Treatment of High-risk Acute T-cell Leukemia / Lymphoma
Brief Title: Phase I Clinical Trial of Autologous CD7-CAR T Cell Therapy for High-risk Acute T-cell Leukemia/lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRYY-IIT-LCYJ-2021-004
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-06

CONDITIONS: T Cell Lymphoma; T-cell Leukemia
MeSH Terms: conditions — Lymphoma, T-Cell; Leukemia, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- chimeric antigen receptor T cell treatment (Experimental)
  Interventions: Biological: chimeric antigen receptor T cell treatment

INTERVENTIONS:
Biological: chimeric antigen receptor T cell treatment — Subjects will be pretreated with chemotherapy prior to infusion of CAR T cells: about 3 days before cells transfusion, the patients who planned to reinfuse CAR T cells were treated with fluorodarabine 30 mg/m2( body surface area) and cyclophosphamide 250 mg/m2( body surface area) for 3 days. Then this study will be using a 3+3 dose escalation approach from dose 1 (DL-1): 5×105 (±20%) to dose 2 (dl-2): 1×106 (±20%). Below the lowest dose was reinfused at the PI's discretion.

SUMMARY:
This is a phase 1 clinical trial of autologous CD7-CAR T cells in the treatment of high-risk acute T-cell leukemia / lymphoma. Twenty subjects will be enrolled. Subjects will be pretreated with chemotherapy prior to infusion of CAR T cells: about 3 days before cells transfusion, the patients who planned to reinfuse CAR T cells were treated with fluorodarabine 30 mg/m2( body surface area) and cyclophosphamide 250 mg/m2( body surface area) for 3 days. Then this study will be using a 3+3 dose escalation approach from dose 1 (DL-1): 5×105 (±20%) to dose 2 (dl-2): 1×106 (±20%). Below the lowest dose was reinfused at the PI's discretion.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Diagnosed as a high-risk acute T-cell leukemia / lymphoma patient with complete remission within 3 months and persistent positive of minimal residual disease, expressing tumor surface antigen CD7
2. Refractory or relapsed T-cell acute lymphoblastic leukemia/lymphoma patients with no blasts in peripheral blood by flow cytometry and suspending anti-neoplastic treatment for more than 2 weeks
3. Male or female, aged 0-70 years
4. No serious allergic constitution
5. Eastern Cooperative Oncology Group (ECOG) performance status (Oken et al., 1982) score 0 to 2
6. Have life expectancy of at least 60 days based on investigator's judgement
7. CD7 positive in bone marrow or peripheral blood or immunohistochemistry
8. Candidates aged 8-70 years need to be sufficiently conscious and able to sign the treatment consent form and voluntary consent form. And Pediatric patients under 8 years old could be recruited after signing an informed consent form by a legal surrogate (Guardian)
9. Minimal residual disease was positive after chemotherapy and there were contraindications of allogeneic hematopoietic stem cell transplantation.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Intracranial hypertension or disorder of consciousness
2. Symptomatic heart failure or severe arrhythmia
3. Symptoms of severe respiratory failure
4. Complicated with other types of malignant tumors
5. Diffuse intravascular coagulation
6. Serum creatinine and / or blood urea nitrogen ≥ 1.5 times of the normal value
7. Suffering from septicemia or other uncontrollable infections
8. Patients with uncontrollable diabetes
9. Severe mental disorders
10. Obvious and active intracranial lesions were detected by cranial magnetic resonance imaging (MRI)
11. Have received organ transplantation (excluding hematopoietic stem cell transplantation);
12. Reproductive-aged female patients with positive blood HCG test
13. Screened to be positive of infection of hepatitis (including hepatitis B and C), AIDS or syphilis

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
DLT rate | 21 days
  The DLT rate to the CAR-T treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Boren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No